CLINICAL TRIAL: NCT00459277
Title: A Multicenter, Placebo-Controlled, Double-Blind, Two-Phase Crossover Study of Nasalfent (Fentanyl Citrate Nasal Spray) in the Treatment of Breakthrough Cancer Pain (BTCP) in Subjects Taking Regular Opioid Therapy
Brief Title: Efficacy & Safety Study of Nasalfent (Fentanyl Citrate Nasal Spray) for Treatment of Breakthrough Cancer Pain in Patients Taking Regular Opioids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Archimedes Development Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CPO43/06/FCNS
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2010-01

CONDITIONS: Cancer Pain
Keywords: Pain; Cancer
MeSH Terms: conditions — Cancer Pain; Pain; Neoplasms | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasalfent, Fentanyl Citrate Nasal Spray (Experimental)
  Interventions: Drug: Fentanyl (Nasalfent, Fentanyl Citrate Nasal Spray)
- Placebo Spray (Placebo Comparator)
  Interventions: Drug: Fentanyl (Nasalfent, Fentanyl Citrate Nasal Spray)

INTERVENTIONS:
Drug: Fentanyl (Nasalfent, Fentanyl Citrate Nasal Spray)

SUMMARY:
Cancer patients taking regular medication for their pain often still have episodes of severe pain that 'break through' despite their background pain treatment. Fentanyl is a strong, short-acting pain killer often used to treat this 'breakthrough' pain. Nasalfent contains fentanyl in a patented drug delivery system called PecSys and is given via a simple nasal spray. This study will test the efficacy and safety of Nasalfent in the treatment of breakthrough cancer pain.

DETAILED DESCRIPTION:
Current treatments for breakthrough cancer pain (BTCP) work too slowly to meet the fast onset of most BTCP episodes, they continue to act longer than the episode of pain lasts and so can have unwanted side effects due to this 'over treatment' of the pain episode. In addition most cancer patients have oral problems which make taking pain relief medication by mouth uncomfortable for the patient. Nasalfent is administered via the nose as a simple spray and can be taken by patients or given by their carers. The nasal route is a common way to administer medication for example in the treatment of migraine or allergy. At any time during the study the patient may take their regular treatment for BTCP should they so wish.

This study will compare the time of onset and degree of pain relief of Nasalfent to that of Placebo. The safety of the two treatments groups (Nasalfent, Placebo) will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give consent
* Women of childbearing potential must have a) negative urine pregnancy test b) not be breast feeding c) agree to practice a reliable form of contraception
* Diagnosis of cancer
* Taking at least 60mg oral morphine or equivalent as 24 hour treatment for cancer-related pain
* Experiencing on average 1 - 4 episodes of breakthrough cancer pain per day usually controlled by rescue pain medication
* Able (or via caregiver)to evaluate and record pain relief, assess medication performance at set times after dosing, record adverse events, record each use of the study drug or rescue medication in a diary
* Able to be up and about for 50% of the day or greater

Exclusion Criteria:

* Intolerance to opioids or fentanyl
* rapidly increasing/uncontrolled pain
* pain that is not cancer related

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2006-12; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Summed pain intensity difference at 30 min | 30 min after dosing

SECONDARY OUTCOMES:
SPID, Pain intensity, Pain intensity difference, Pain relief and Total pain relief | Various timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Russell K Portenoy, MD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Taylor D, Galan V, Weinstein SM, Reyes E, Pupo-Araya AR, Rauck R; Fentanyl Pectin Nasal Spray 043 Study Group. Fentanyl pectin nasal spray in breakthrough cancer pain. J Support Oncol. 2010 Jul-Aug;8(4):184-90. PMID 20822038